CLINICAL TRIAL: NCT01405456
Title: Randomized Placebo-controlled Trial to Investigate the Effects of Eplerenone in Patients With HIV-associated Abdominal Fat Accumulation
Brief Title: Eplerenone in HIV Associated Abdominal Fat Accumulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010P002095
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: HIV
Keywords: HIV-infection; eplerenone; aldosterone; visceral fat; lipodystrophy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Lipodystrophy | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eplerenone and Lifestyle (Experimental): First 6 months: eplerenone 50mg daily along with lifestyle modification (counseling regarding lifestyle and diet, as well as following healthy activity guidelines) Second 6 months: same (eplerenone open label during second 6 months)
  Interventions: Drug: Eplerenone and lifestyle
- Placebo and Lifestyle (Placebo Comparator): First 6 months: placebo pill daily along with lifestyle modification (counseling regarding lifestyle and diet, as well as following healthy activity guidelines) Second 6 months: eplerenone (open label) 50mg daily along with continued lifestyle modification
  Interventions: Other: placebo and lifestyle

INTERVENTIONS:
Drug: Eplerenone and lifestyle — eplerenone 50mg by mouth daily as well as lifestyle counseling
  Arms: Eplerenone and Lifestyle
Other: placebo and lifestyle — placebo pill daily and lifestyle counseling
  Arms: Placebo and Lifestyle

SUMMARY:
The purpose of this study is to test the effects of a drug, eplerenone, along with lifestyle modification to affect sugar metabolism, body fat distribution, and cardiovascular health in HIV-infected individuals. In non-HIV-infected individuals, recent data has shown that aldosterone, a hormone that regulates salt and water balance, is increased in association with increased belly fat and decreased insulin sensitivity. In HIV-infected individuals, aldosterone appears to be higher in individuals with increased belly fat, and increased aldosterone appears to be strongly associated with impaired sugar metabolism. In this study, the investigators will test the effects of eplerenone, which is a medication that blocks the actions of aldosterone, along with lifestyle modification. The investigators hypothesize that eplerenone may improve sugar metabolism, improve markers of cardiovascular health, and reduce fat accumulation in liver and muscle.

DETAILED DESCRIPTION:
The study is 12 months long, with two phases. In the initial, 6-month phase, volunteers are randomly assigned to receive either eplerenone or placebo (an inactive pill). In addition, all volunteers will receive counseling about healthy diet and lifestyle, and will be asked to follow guidelines for a healthy level of physical activity. In the second 6-months of the study, all volunteers will continue to receive lifestyle modification and all will receive eplerenone.

ELIGIBILITY:
Inclusion Criteria:

1. Increased waist circumference based on NCEP guidelines (>102cm in men and >88cm in women) and impaired glucose tolerance (either IFG > 100 mg/dL but < 126 mg/dL or 2hr glucose > 140 mg/dl but < 200 mg/dL, or fasting insulin >12 uIU/mL)
2. HIV positive for 5y and on a stable ART regimen for at least 12 months
3. Age ≥ 30 and ≤ 65 years of age

Exclusion Criteria:

1. ACE Inhibitor, ARB, verapamil, or spironolactone
2. Potassium supplementation
3. Estimated GFR<60, creatinine > 1.5 mg/dL
4. Serum K > 5.5 mEq/L, ALT > 2.5 times the upper limit of normal, Hgb < 11g/dL
5. Uncontrolled hypertension (SBP ≥ 160 or DBP ≥ 100)
6. Current or prior steroid use within past 6 months
7. Known history of diabetes mellitus or current use of anti-diabetic medications
8. Concomitant use of full dose ritonavir, nelfinavir, clarithromycin and other strong inhibitors of CYP34A
9. Use of St. John's Wart (CYP3A4 inducer)
10. Pregnant or actively seeking pregnancy, breastfeeding
11. For women: Pregnant or actively seeking pregnancy, breastfeeding, failure to use an acceptable non-hormonal form of birth control, including abstinence, barrier contraceptives, or non-hormonal IUD.
12. Estrogen or progestational derivative use within 3 months
13. Testosterone use for non-physiologic purposes, or physiologic testosterone replacement for < 3 months.
14. Current growth hormone or growth hormone releasing hormone use
15. Current viral, bacterial or other infections (excluding HIV)
16. Current active substance abuse
17. Patients with a significant history of cardiovascular disease, including prior MI or stroke

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-01; Primary Completion 2017-05-03 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Srinivasa S, deFilippi C, Fitch KV, Iyengar S, Shen G, Burdo TH, Walpert AR, Thomas TS, Adler GK, Grinspoon SK. Evaluation of Mineralocorticoid Receptor Antagonism on Changes in NT-proBNP Among Persons With HIV. J Endocr Soc. 2021 Nov 19;6(1):bvab175. doi: 10.1210/jendso/bvab175. eCollection 2022 Jan 1. PMID 34909518
- [Derived] Srinivasa S, Fitch KV, Wong K, O'Malley TK, Maehler P, Branch KL, Looby SE, Burdo TH, Martinez-Salazar EL, Torriani M, Lyons SH, Weiss J, Feldpausch M, Stanley TL, Adler GK, Grinspoon SK. Randomized, Placebo-Controlled Trial to Evaluate Effects of Eplerenone on Metabolic and Inflammatory Indices in HIV. J Clin Endocrinol Metab. 2018 Jun 1;103(6):2376-2384. doi: 10.1210/jc.2018-00330. PMID 29659888

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eplerenone and Lifestyle | Placebo and Lifestyle
Started | 25 | 21
Completed | 22 | 20
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eplerenone and Lifestyle | Placebo and Lifestyle | Total
Number analyzed (Participants) | 25 | 21 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (6) | 52 (6) | 51 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 15 | 15 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 11 | 20
  White | 15 | 9 | 24
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 21 | 46
Insulin Stimulated Glucose Uptake [Median (Inter-Quartile Range); unit: mg/min per μIU/ml] — Insulin stimulated glucose uptake at steady state using the euglycemic hyperinsulinemic clamp technique normalized to insulin and lean body mass. Population: Endpoint could not be obtained. Subject was unable to complete the procedure.
  mg/min per μIU/ml
    number analyzed (Participants) | 24 | 21 | 45
    (all) | 7.26 [5.74 to 9.55] | 7.52 [5.12 to 10.43] | 7.44 [5.64 to 9.87]
Visceral Adipose Tissue [Median (Inter-Quartile Range); unit: cm^2] — Abdominal visceral fat obtained by MRI. Population: Endpoint could not be obtained. Subjects could could not complete the procedure.
  cm^2
    number analyzed (Participants) | 23 | 21 | 44
    (all) | 215 [154 to 324] | 241 [147 to 295] | 230 [154 to 308]
Liver Fat [Median (Inter-Quartile Range); unit: percentage of intrahepatic lipid] — Intrahepatic lipid obtained by MRS. Population: Endpoint could not be obtained. Subjects could not complete the procedure.
  percentage of intrahepatic lipid
    number analyzed (Participants) | 22 | 21 | 43
    (all) | 5 [3 to 12] | 5 [2 to 12] | 5 [3 to 12]
Intramyocellular Lipid [Median (Inter-Quartile Range); unit: percentage of intramyocellular lipid] — Intramyocellular lipid of the tibialis anterior muscle obtained by MRS. Population: Endpoint could not be obtained. Subjects could not complete the procedure.
  percentage of intramyocellular lipid
    number analyzed (Participants) | 24 | 21 | 45
    (all) | 0.5 [0.2 to 0.6] | 0.3 [0.2 to 0.5] | 0.4 [0.2 to 0.5]
Flow Mediated Vasodilation [Median (Inter-Quartile Range); unit: percentage of maximum change] — Flow mediated vasodilation obtained at the brachial artery. Population: Endpoint could not be obtained. Studies were of poor quality and data could not be analyzed.
  percentage of maximum change
    number analyzed (Participants) | 24 | 19 | 43
    (all) | 13.0 [9.7 to 19.3] | 13.4 [10.8 to 17.6] | 13.0 [10.7 to 17.6]
Potassium [Mean (Standard Deviation); unit: mEq/L] | 4.1 (0.2) | 4.0 (0.2) | 4.1 (0.2)
Hemoglobin A1c [Median (Inter-Quartile Range); unit: percentage] | 5.7 [5.5 to 6.0] | 5.8 [5.3 to 6.1] | 5.7 [5.5 to 6.0]
C-reactive Protein [Median (Inter-Quartile Range); unit: mg/L] — Population: Endpoint could not be evaluated. Sufficient sample was not obtained.
  mg/L
    number analyzed (Participants) | 24 | 21 | 45
    (all) | 3.3 [1.2 to 9.4] | 3.7 [1.6 to 9.8] | 3.4 [1.3 to 9.6]
Plasminogen Activator Inhibitor 1 [Mean (Standard Deviation); unit: ng/mL] — Population: Endpoint could not be obtained. Sufficient sample was not obtained.
  ng/mL
    number analyzed (Participants) | 24 | 21 | 45
    (all) | 36.7 (18.3) | 37.0 (18.7) | 36.9 (18.3)
Adiponectin [Median (Inter-Quartile Range); unit: pg/mL] — Population: Endpoint could not be evaluated. Sufficient sample was not obtained.
  pg/mL
    number analyzed (Participants) | 24 | 21 | 45
    (all) | 4016 [3439 to 5360] | 4673 [3302 to 6042] | 4527 [3373 to 5484]
Markers of Systemic Inflammation [Median (Inter-Quartile Range); unit: pg/mL] — IL-6 Population: Endpoint could not be evaluated. Sufficient sample was not obtained.
  pg/mL
    number analyzed (Participants) | 24 | 21 | 45
    (all) | 10.2 [5.2 to 19.8] | 7.9 [6.1 to 18.3] | 9.1 [5.9 to 19.3]
Markers of Immune Activation [Mean (Standard Deviation); unit: pg/mL] — MCP-1 Population: Endpoint could not be evaluated. Sufficient sample was not obtained.
  pg/mL
    number analyzed (Participants) | 24 | 21 | 45
    (all) | 205 (78) | 191 (51) | 198 (66)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Stimulated Glucose Uptake
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: mg/min per μIU/ml
Arm/Group | Eplerenone and Lifestyle | Placebo and Lifestyle
Number analyzed (Participants) | 21 | 20
mg/min per μIU/ml | 7.70 [5.01 to 8.36] | 8.58 [5.76 to 12.30]
Statistical Analysis 1: Comparison: Eplerenone and Lifestyle vs Placebo and Lifestyle; Change in Insulin Stimulated Glucose Uptake measured during euglycemic hyperinsulinemic clamp procedure from baseline to 6 months; Test type: Superiority; p = 0.71, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Visceral Adipose Tissue
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: cm^2
Arm/Group | Eplerenone and Lifestyle | Placebo and Lifestyle
Number analyzed (Participants) | 20 | 20
cm^2 | 231 [145 to 327] | 233 [142 to 318]
Statistical Analysis 1: Comparison: Eplerenone and Lifestyle vs Placebo and Lifestyle; Change in Visceral Adipose Tissue area as measured by magnetic resonance imaging of the abdomen from baseline to 6 months; Test type: Superiority; p = 0.42, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Liver Fat
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: percentage of intrahepatic lipid
Arm/Group | Eplerenone and Lifestyle | Placebo and Lifestyle
Number analyzed (Participants) | 19 | 18
percentage of intrahepatic lipid | 6 [3 to 13] | 4 [2 to 9]
Statistical Analysis 1: Comparison: Eplerenone and Lifestyle vs Placebo and Lifestyle; Change in Liver Fat (Intrahepatic Lipid) as measured by magnetic resonance spectroscopy from baseline to 6 months; Test type: Superiority; p = 0.51, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Intramyocellular Lipid
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: percentage of intramyocellular lipid
Arm/Group | Eplerenone and Lifestyle | Placebo and Lifestyle
Number analyzed (Participants) | 20 | 20
percentage of intramyocellular lipid | 0.4 [0.2 to 0.6] | 0.4 [0.3 to 0.4]
Statistical Analysis 1: Comparison: Eplerenone and Lifestyle vs Placebo and Lifestyle; Change in Intramyocellular Lipid of calf muscles as measured by magnetic resonance spectroscopy from baseline to 6 months; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Flow Mediated Vasodilation
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: percentage of maximum change
Arm/Group | Eplerenone and Lifestyle | Placebo and Lifestyle
Number analyzed (Participants) | 20 | 17
percentage of maximum change | 15.3 [7.7 to 17.3] | 9.6 [6.9 to 20.4]
Statistical Analysis 1: Comparison: Eplerenone and Lifestyle vs Placebo and Lifestyle; Change in Flow Mediated Vasodilation (maximum percentage) from baseline to 6 months; Test type: Superiority; p = 0.44, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Potassium
Time Frame: 6 months
Measure: Mean (Standard Error); unit: mEq/L
Arm/Group | Eplerenone and Lifestyle | Placebo and Lifestyle
Number analyzed (Participants) | 22 | 20
mEq/L | 4.2 (0.1) | 4.2 (0.0)
Statistical Analysis 1: Comparison: Eplerenone and Lifestyle vs Placebo and Lifestyle; Mean serum measurements of Potassium; Test type: Superiority; p = 0.07, t-test, 2 sided

7. Secondary Outcome: Hemoglobin A1c
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Eplerenone and Lifestyle | Placebo and Lifestyle
Number analyzed (Participants) | 22 | 20
percentage | 5.7 [5.4 to 6.0] | 5.8 [5.4 to 5.9]
Statistical Analysis 1: Comparison: Eplerenone and Lifestyle vs Placebo and Lifestyle; Change in Hemoglobin A1c from baseline to 6 months; Test type: Superiority; p = 0.70, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: C-Reactive Protein
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Eplerenone and Lifestyle | Placebo and Lifestyle
Number analyzed (Participants) | 21 | 18
mg/L | 2.8 [1.7 to 5.8] | 2.8 [0.9 to 10.3]
Statistical Analysis 1: Comparison: Eplerenone and Lifestyle vs Placebo and Lifestyle; Change in C-Reactive Protein from baseline to 6 months; Test type: Superiority; p = 0.10, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Plasminogen Activator Inhibitor 1
Time Frame: 6 months
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Eplerenone and Lifestyle | Placebo and Lifestyle
Number analyzed (Participants) | 21 | 18
ng/mL | 35 (3) | 35 (3)
Statistical Analysis 1: Comparison: Eplerenone and Lifestyle vs Placebo and Lifestyle; Change in Plasminogen Activator Inhibitor 1 from baseline to 6 months; Test type: Superiority; p = 0.37, t-test, 2 sided

10. Secondary Outcome: Adiponectin
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Eplerenone and Lifestyle | Placebo and Lifestyle
Number analyzed (Participants) | 21 | 18
pg/mL | 4015 [2926 to 5588] | 4014 [3213 to 6012]
Statistical Analysis 1: Comparison: Eplerenone and Lifestyle vs Placebo and Lifestyle; Change in Adiponectin from baseline to 6 months; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Markers of Systemic Inflammation
Description: IL-6
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Eplerenone and Lifestyle | Placebo and Lifestyle
Number analyzed (Participants) | 21 | 17
pg/mL | 9.8 [4.8 to 16.6] | 8.9 [6.3 to 27.8]
Statistical Analysis 1: Comparison: Eplerenone and Lifestyle vs Placebo and Lifestyle; Change in IL-6 from baseline to 6 months; Test type: Superiority; p = 0.10, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Markers of Immune Activation
Description: MCP-1
Time Frame: 6 months
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Eplerenone and Lifestyle | Placebo and Lifestyle
Number analyzed (Participants) | 21 | 18
pg/mL | 205 (19) | 210 (17)
Statistical Analysis 1: Comparison: Eplerenone and Lifestyle vs Placebo and Lifestyle; Change in MCP-1 from baseline to 6 months; Test type: Superiority; p = 0.04, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Eplerenone and Lifestyle | Placebo and Lifestyle
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/21
Other Adverse Events (participants affected / at risk) | 13/25 | 11/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eplerenone and Lifestyle (N=25) | Placebo and Lifestyle (N=21)
Elevated Creatinine (Renal and urinary disorders) | 1 (1) | 1 (1)
Dizziness (Cardiac disorders) | 1 (1) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 2 (2)
Headache (General disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal Bleed (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Other Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Symptoms (Renal and urinary disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Mood Symptoms (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT01405456/Prot_SAP_001.pdf